CLINICAL TRIAL: NCT04719650
Title: The Pharmacokinetics and Pharmacodynamics Study of Intravenous Zoledronic Acid in Chinese Subjects With Low Bone Mass or Osteoporosis: a Randomized Placebo-controlled Trail
Brief Title: Clinical Pharmacokinetics and Pharmacodynamics Study of Different Doses of Zoledronic Acid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2020427
Record Dates: First submitted 2021-01-07; First posted 2021-01-22 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-01

CONDITIONS: Postmenopausal Osteoporosis
Keywords: zoledronic acid; pharmacokinetic; pharmacodynamic; Chinese osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- zoledronic acid 1mg (Experimental): Add 20 mL of Zoledronic acid injection (100mL : 5mg) with 80 mL of normal saline to 100 mL. Infusion 20 minutes with constant speed. Administration only once.
  Interventions: Drug: Zoledronic Acid Injection
- zoledronic acid 2.5mg (Experimental): Add 50 mL of Zoledronic acid injection (100mL : 5mg) with 50 mL of normal saline to 100 mL. Infusion 20 minutes with constant speed. Administration only once.
  Interventions: Drug: Zoledronic Acid Injection
- zoledronic acid 5mg (Experimental): Infusion 100 mL of Zoledronic acid injection (100mL : 5mg) with constant speed in 20 minutes. Administration only once.
  Interventions: Drug: Zoledronic Acid Injection
- placebo (Placebo Comparator): Infusion 100 mL of normal saline with constant speed in 20 minutes. Administration only once.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid Injection — Infusion 1mg zoledronic acid once.
  Other Names: Yigu
  Arms: zoledronic acid 1mg
Drug: Zoledronic Acid Injection — Infusion 2.5mg zoledronic acid once.
  Other Names: Yigu
  Arms: zoledronic acid 2.5mg
Drug: Zoledronic Acid Injection — Infusion 5mg zoledronic acid once.
  Other Names: Yigu
  Arms: zoledronic acid 5mg
Drug: Placebo — Infusion normal saline once.
  Other Names: Yigu Placebo
  Arms: placebo

SUMMARY:
The recommended dosing regimen of zoledronic acid in Chinese osteoporosis patients is completely in accordance with the one of 5 mg per year abroad that based on the dosing regimen in Paget's disease. This dosing regimen lacks the actual supportive clinical data of Chinese patients. In addition, the overall incidence of acute phase response, the main adverse event after the first infusion, in Chinese patients is higher than that in Caucasian patients population. Moreover, the results of the similar drug clinical study in the Japanese patients shown that the purpose of effective treatment for osteoporosis could be achieved with half of the dosage in Caucasian population. Thus, it could be inferred from these that the dosing regimen of zoledronic acid might be inappropriate in Chinese osteoporosis patients. Therefore, the main purpose of this clinical trail is to compare the zoledronic acid pharmacokinetic and pharmacodynamic characteristic of different doses in Chinese postmenopausal subjects with low bone mass or osteoporosis and explore the best dosing regimen in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese postmenopausal women
2. Aged between 60 and 70.
3. Bone mineral density (BMD) values of less than 1 standard deviations (SD) below the normal adult mean.
4. Willing to participate in this study.

Exclusion Criteria:

1. Hypersensitivity to zoledronic acid or other bisphosphonate or zoledronic acid formulation (excipients).
2. Secondary osteoporosis.
3. Receiving the following drugs that affect bone metabolism prior to randomization:

(1) intravenous biphosphonates or denosumab. (2) oral biphosphonates, parathyroid hormone or its analogues, strontium, or fluoride within 12 months.

(3) glucocorticoid, steroids, immunosuppressive agents, calcitonin, calcitriol or its analogues, thiazides diuretics, long-acting estrogen/progesterone, or statins within 3 months.

4. Combine other diseases affect bone metabolism: osteogenesis imperfecta, hyperthyroidism, malignant tumors, Paget's disease, rheumatoid arthritis, osteomalacia, osteopetrosis, ankylosing spondylitis, liver failure, or renal failure.

5. Hyperthyroidism or hypothyroidism during screening.

6. Treatment with any investigational drug within the past 3 months.

7. Creatinine clearance < 35 mL/min.

8. 25(OH)D level< 20 ng/mL.

9. Serum calcium level < 2.0 mmol/L (8 mg/dL), or >2.8 mmol/L (11.0 mg/dL).

10. Fever, severe infections, severe injuries, or major surgical operation within 30 days.

11. ECG corrected QT interval (QTc) > 480 ms.

12. Pending invasive dental procedure or in progress.

13. History of smoking within 6 months.

14. Diabetes with fasting blood glucose ≥ 7.0 mmol/L, or glycated hemoglobin (HbA1c) >6.3%.

15. History of drug or alcohol abuse.

16. History of stroke, cerebral ischemic stroke, or cerebral hemorrhage.

17. Any physiological or medical condition which, in the opinion of the investigator, would preclude the participant from this trail.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of Zoledronic acid | Predose, 30 minutes, 2 hours, 24 hours, day 7, day 29, 3 months, 6 months, 12 months, 24 months, and 36 months post dose
  Zoledronic acid concentration in plasma and urine.
Maximum concentration of Zoledronic acid | 0-36 months
  The observed maximum concentration following administration (Cmax) in plasma after zoledronic acid infusion.
Time to reach maximum concentration of Zoledronic acid | 0-36 months
  The time to reach the maximum concentration after administration (Tmax) in plasma after zoledronic acid infusion.
AUC of Zoledronic acid | 0-36 months
  The area under the concentration-time curve (AUC) in plasma after zoledronic acid infusion.
terminal half-life of Zoledronic acid | 0-36 months
  The terminal half-life (t1/2) of zoledronic acid after administration.
apparent clearance of Zoledronic acid | 0-36 months
  The apparent clearance (CL/F) of zoledronic acid after administration.
apparent volume of distribution of Zoledronic acid | 0-36 months
  The apparent volume of distribution of zoledronic acid after administration.
Concentration of bone turnover markers | 0-36 months
  Concentration-time profile of procollagen type 1 N-propeptide (P1NP), bone-specific alkaline phosphatase (ALP), osteocalcin (OCN), C-telopeptide (CTx), and tartrate-resistant acid phosphatase 5b (TRACP-5b) with unit of ng/mL.
Concentration of 25(OH)D and FGF23 | 0-36 months
  Concentration determination of 25(OH)D and fibroblast growth factor 23 (FGF23) with unit of ng/mL
PTH concentration determination | 0-36 months
  Assessment of the profile of parathyroid hormone (PTH)
Serum sclerostin concentration determination | 0-36 months
  Concentration-time profile of sclerostin (SOST) after zoledronic acid infusion.
Pharmacodynamic of zoledronic acid | 0-36 months
  Assessment of lipid metabolism markers, such as low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol, and triglycerides.
Pharmacodynamic of zoledronic acid | 0-36 months
  Assessment of fibroblast growth factor 19 (FGF19).
Pharmacodynamic of zoledronic acid | 0-36 months
  Assessment of total bile acid.
Pharmacodynamic of zoledronic acid | 0-36 months
  Assessment of bone mineral density at the lumbar spine, neck of femur, and total hip.
Change of immune indicator | 0-36 months
  Changes in white blood cells(WBC)
Change of immune indicator | 0-36 months
  Changes in C reaction protein (CRP)
Change of immune indicator | 0-36 months
  Changes in interferon-γ (IFN-γ)
Change of immune indicator | 0-36 months
  Changes in interleukin-6 (IL-6)
Change of immune indicator | 0-36 months
  Changes in γδT cells activation

SECONDARY OUTCOMES:
Incidence of adverse event | 0-36 months
  The occurrence time and severity of fracture. The occurrence time and severity of acute phase response. The occurrence time and severity of other adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, M.D.; Ph. D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Shiraki M, Fukunaga M, Kushida K, Kishimoto H, Taketani Y, Minaguchi H, Inoue T, Morita R, Morii H, Yamamoto K, Ohashi Y, Orimo H. A double-blind dose-ranging study of risedronate in Japanese patients with osteoporosis (a study by the Risedronate Late Phase II Research Group). Osteoporos Int. 2003 May;14(3):225-34. doi: 10.1007/s00198-002-1369-9. Epub 2003 Apr 10. PMID 12730746
- [Background] Ding Y, Zeng JC, Yin F, Zhang CL, Zhang Y, Li SX, Liu X, Zhang C, Xue QY, Lin H, Pei FX. Multicenter Study on Observation of Acute-phase Responses After Infusion of Zoledronic Acid 5 mg in Chinese Women with Postmenopausal Osteoporosis. Orthop Surg. 2017 Aug;9(3):284-289. doi: 10.1111/os.12338. PMID 28960821